CLINICAL TRIAL: NCT02466191
Title: Treatment of Pendular Nystagmus With Gabapentin and Memantine in Patients With Oculopalatal Tremor: a Controled Open-label Study
Brief Title: Treatment of Pendular Nystagmus in OPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL14_0438; 2014-005548-17 (EudraCT Number)
Record Dates: First submitted 2015-05-22; First posted 2015-06-09 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pendular Nystagmus; Oculopalatal Tremor
Keywords: nystagmus; pharmacological trial; multiple sclerosis; oscillopsia
MeSH Terms: conditions — Nystagmus, Pathologic; Multiple Sclerosis | interventions — Memantine; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- memantine first (Experimental): Patients will be randomly assigned to start on either memantine or gabapentin. For tolerance reasons, each treatment begins with a progressive increasing dose and stops with a progressive decreasing dose. The duration of the period of last dose (8 to 11 days) will be chosen according to the investigator's availability to organize post-tests.
  Interventions: Drug: Memantine
- gabapentin first (Experimental): Patients will be randomly assigned to start on either memantine or gabapentin. For tolerance reasons, each treatment begins with a progressive increasing dose and stops with a progressive decreasing dose. The duration of the period of last dose (8 to 11 days) will be chosen according to the investigator's availability to organize post-tests.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Memantine
  Arms: memantine first
Drug: Gabapentin
  Arms: gabapentin first

SUMMARY:
Pendular nystagmus corresponds to an enduring to and fro eye oscillation without resetting quick phases. The most common causes of acquired pendular nystagmus (APN) are multiple sclerosis (MS) and focal brainstem lesions (oculopalatal tremor, OPT). Based on pathophysiological hypothesis, pharmacological treatments of acquired nystagmus have been thoroughly proposed over different publications of cases, series, reviews or expert opinions. Acquired pendular nystagmus underwent the most rigorous treatment trials, leading to the proposal of gabapentin or memantine as valuable drugs. Whether gabapentin and memantine are effective in APN associated with OPT remains unclear, since none of the previous studies has evaluated the effect of these medications in a group of OPT patients. However, this is an important issue in prospect to a clinical use of these medications. In the current study, the investigators aim is to evaluate the effect of gabapentin and memantine on the mean velocity, amplitude and frequency of pendular nystagmus, as well as on visual acuity and vision-specific health-related quality of life score, in a group of OPT patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of oculopalatal tremor (OPT), following a focal brainstem lesion.
* All patients may present a chronic acquired pendular nystagmus due to OPT, observed over a period of 6 months.
* All patients will be informed about the design and purpose of the study, and all will give their informed, written consent to the protocol, which may have been approved by the local ethics committee.
* Age: above 18
* Able to understand the instructions
* Having a health coverage
* Able to sit down for 1 hour
* Stable dosage of previous medications (beginning 3 weeks previously and terminating at the end of the trial duration), except gabapentin or memantine.
* For women: efficient contraception during the experimental time and in the two month following treatment withdrawal.

Exclusion Criteria:

* Ophthalmological

  * Other ophthalmological disorder that could impair corrected visual acuity (Maculopathy, Retinopathy…)
* Neurological

  * Ongoing seizure
  * Severe handicap that does not allow sitting down position for 1 hour
* Suicidal behavior or risk
* Treatment

  * Under memantine or gabapentin medication (these medications should have been stopped for at least 1 week for gabapentin and 3 weeks for memantine)
  * Under morphine, N-methyl-D-aspartate such as amantadine, ketamine or dextromethorphan
  * Steroid medication for a current relapse (beginning 3 weeks previously and terminating at the end of the trial duration
  * Known hypersensitivity to memantine or gabapentin
* General

  * Unstable medical state
  * Patient with a galactose intolerance, a lapp lactase deficiency or glucose-galactose malabsorption
  * Moderate renal failure (creatinine clearance < 50 mL/min on bioassay dated from less than one month)
  * Recent heart infarction (<3months)
  * Unstable congestive heart insufficiency
  * Unstable arterial hypertension
  * Leucopenia (<2500/mm3)
  * Transaminase increase (>5 time normal values)
* Pregnancy (on questioning)
* Tutelage or any legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Velocity, amplitude and frequency of nystagmus using eye movement recording | at Day 17-21
Velocity, amplitude and frequency of nystagmus using eye movement recording | at Day 34-42
Velocity, amplitude and frequency of nystagmus using eye movement recording | at Day 64-79
Velocity, amplitude and frequency of nystagmus using eye movement recording | at Day 81-100

SECONDARY OUTCOMES:
Functional score on questioning as measured by the 25-Item National Eye Institute Visual Function Questionnaire | at Day 17-21
Functional score on questioning as measured by the 25-Item National Eye Institute Visual Function Questionnaire | at Day 34-42
Functional score on questioning as measured by the 25-Item National Eye Institute Visual Function Questionnaire | at Day 64-79
Functional score on questioning as measured by the 25-Item National Eye Institute Visual Function Questionnaire | at Day 81-100
subjective measure of oscillopsia | at Day 17-21
subjective measure of oscillopsia | at Day 34-42
subjective measure of oscillopsia | at Day 64-79
subjective measure of oscillopsia | at Day 81-100
far visual acuity as measured by monocularly and binocularly direction and amplitude (measures in degrees) of their oscillopsia while viewing, with best correction, a stationary target at far (5 m) and near (57 cm) location. | at Day 17-21
far visual acuity as measured by monocularly and binocularly direction and amplitude (measures in degrees) of their oscillopsia while viewing, with best correction, a stationary target at far (5 m) and near (57 cm) location. | at Day 34-42
far visual acuity as measured by monocularly and binocularly direction and amplitude (measures in degrees) of their oscillopsia while viewing, with best correction, a stationary target at far (5 m) and near (57 cm) location. | at Day 64-79
far visual acuity as measured by monocularly and binocularly direction and amplitude (measures in degrees) of their oscillopsia while viewing, with best correction, a stationary target at far (5 m) and near (57 cm) location. | at Day 81-100

CONTACTS AND LOCATIONS:
Overall Officials: Caroline TILIKETE, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Background] Nerrant E, Abouaf L, Pollet-Villard F, Vie AL, Vukusic S, Berthiller J, Colombet B, Vighetto A, Tilikete C. Gabapentin and Memantine for Treatment of Acquired Pendular Nystagmus: Effects on Visual Outcomes. J Neuroophthalmol. 2020 Jun;40(2):198-206. doi: 10.1097/WNO.0000000000000807. PMID 31169568